CLINICAL TRIAL: NCT01066936
Title: Bone Density by Dual Energy X-ray Absorptiometry (DEXA) Following Total Hip Arthroplasty With the "Short Mini Stem"
Brief Title: Mini Stem DEXA (Dual Energy X-ray Absorptiometry)
Acronym: MISDexa
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2090SMFH131
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the bone ingrowth after implantation of the study device. This study will also document any device-related surgical complications or adverse radiographic observations. Improvement in pain, function, and health economic data will be compared with improvements documented with other joint systems.

DETAILED DESCRIPTION:
The purpose of the current investigation is to assess the bone ingrowth after implantation with a modular, short hip stem using Dual Energy X-ray Absorptiometry (DEXA). The intended use of this product is for patients with non-inflammatory and inflammatory degenerative joint disease who require a primary total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patient has hip disease that requires a total hip arthroplasty.
* Patient is willing to consent to participate in the study.
* Patient plans to be available for the study duration.
* Patient is in stable health and is free of or treated and stabilized for cardiac, pulmonary, hematological, or other conditions that would pose excessive operative risk.

Exclusion Criteria:

* Patient known to have insufficient bone stock.
* Patient has had major non-arthroscopic surgery to the study hip.
* Patient has physical, emotional or neurological conditions that would compromise the patient's compliance with postoperative rehabilitation and follow-up.
* Patient has a known sensitivity to materials in the device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The purpose of this investigation is to assess the bone growth after implantation with a modular, short hip stem using Dual Energy X-ray Absorptiometry (DEXA). The intended use of this product is for patients with non-inflammatory and inflammatory degenerative joint disease who require a total hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-09-14 (Actual); Primary Completion 2016-04-18 (Actual); Study Completion 2016-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve McMahon, MD, Principal Investigator — Malabar Orthopaedic Clinic; Beate Hanson, MD, PhD, Study Chair — Vice Presidient, Global Clinical Strategy
Locations (1):
- Malabar Orthopaedic Clinic, Windsor, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by 1 investigator in 1 country from 14 Sep 2009 to 18 Apr 2016.
Pre-assignment Details: A total of 22 subjects were screened, with 20 subjects enrolled and had surgery/MIS implanted.
Units Other Than Participants: hips
Groups:
- MIS (Mini Stem) Stem: Patients with non-inflammatory and inflammatory degenerative joint disease (DJD) who required a primary total hip replacement (THR) and had the MIS femoral stem/modular neck implanted. There was no assignment of study treatment: all subjects had implantation of the MIS femoral stem/modular neck during total hip arthroplasty (THA).
Period: Overall Study
Arm/Group | MIS (Mini Stem) Stem
Started | 20; 20 hips
Completed | 10; 10 hips
Not Completed | 10; 10 hips
Not completed — Death | 2
Not completed — Device revised/removed | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- MIS Stem: Patients with non-inflammatory and inflammatory degenerative joint disease (DJD) who required a primary total hip replacement (THR) and had the MIS femoral stem/modular neck implanted. All subjects had implantation of the MIS femoral stem/modular neck during THA. DEXA was used to assess the bone ingrowth and detect significant alterations in skeletal structure that may not be visible during routine clinical assessment.
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 19
  European | 1
Region of Enrollment [Number; unit: participants]
  Australia | 20
Height [Mean (Standard Deviation); unit: cm] | 170.2 (7.39)
Weight [Mean (Standard Deviation); unit: kg] | 90.8 (12.39)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (3.69)
Primary Diagnosis Charnley Classification [Count of Participants; unit: Participants]
  Avascular necrosis: B1 Bilateral Hip Joint Disease | 1
  Osteoarthritis: A Unilateral Hip Joint Disease | 14
  Osteoarthritis: B1 Bilateral Hip Joint Disease | 4
  Rheumatoid arthritis:C1 Multi-joint arthroplasties | 1

OUTCOME MEASURES:

1. Primary Outcome: DEXA Analysis of BMD at Preoperative Visit
Description: DEXA=Dual Energy X-Ray Absorptiometry; BMD=Bone Mineral Density; The proximal femur was divided into 7 regions relative to the length of the stem. Lateral portions = region 1, region 2 and region 3; The entire bone mass immediately distal to the stem tip = region 4; Medial portions = region 5, region 6, and region 7. Mean BMD was calculated for each femoral region. BMD values were adjusted peri-prosthetically to account for stem area.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: g/cm^2
Groups:
- MIS Stem: Patients with non-inflammatory and inflammatory degenerative joint disease (DJD) who required a primary total hip replacement (THR) and had the MIS femoral stem/modular neck implanted.
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
g/cm^2
  Femoral Region 1 | 0.8 (0.22)
  Femoral Region 2 | 1.0 (0.25)
  Femoral Region 3 | 1.6 (0.31)
  Femoral Region 4 | 2.0 (0.32)
  Femoral Region 5 | 1.8 (0.33)
  Femoral Region 6 | 1.3 (0.29)
  Femoral Region 7 | 1.4 (0.31)

2. Primary Outcome: DEXA Analysis of BMD at 3 Months
Description: as for outcome 1
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: g/cm^2
Groups:
- Study Population: Patients with non-inflammatory and inflammatory degenerative joint disease (DJD) who required a primary total hip replacement (THR) and had the MIS femoral stem/modular neck implanted.
Arm/Group | Study Population
Number analyzed (Participants) | 20
g/cm^2
  Femoral Region 1 | 0.8 (0.18)
  Femoral Region 2 | 1.3 (0.26)
  Femoral Region 3 | 2.1 (0.39)
  Femoral Region 4 | 1.9 (0.27)
  Femoral Region 5 | 1.9 (0.27)
  Femoral Region 6 | 1.5 (0.32)
  Femoral Region 7 | 1.3 (0.27)

3. Primary Outcome: DEXA Analysis of BMD at 6 Months
Description: as for outcome 1
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Study Population
Number analyzed (Participants) | 20
g/cm^2
  Femoral Region 1 | 0.8 (0.19)
  Femoral Region 2 | 1.3 (0.31)
  Femoral Region 3 | 2.1 (0.38)
  Femoral Region 4 | 1.9 (0.30)
  Femoral Region 5 | 2.0 (0.28)
  Femoral Region 6 | 1.6 (0.30)
  Femoral Region 7 | 1.2 (0.35)

4. Primary Outcome: DEXA Analysis of BMD at 1 Year
Description: as for outcome 1
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Study Population
Number analyzed (Participants) | 20
g/cm^2
  Femoral Region 1 | 0.8 (0.20)
  Femoral Region 2 | 1.3 (0.29)
  Femoral Region 3 | 2.1 (0.41)
  Femoral Region 4 | 1.9 (0.30)
  Femoral Region 5 | 1.9 (0.31)
  Femoral Region 6 | 1.6 (0.37)
  Femoral Region 7 | 1.3 (0.30)

5. Primary Outcome: DEXA Analysis of BMD at 2 Years
Description: as for outcome 1
Time Frame: 2 Year
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Study Population
Number analyzed (Participants) | 19
g/cm^2
  Femoral Region 1 | 0.8 (0.21)
  Femoral Region 2 | 1.3 (0.33)
  Femoral Region 3 | 2.2 (0.31)
  Femoral Region 4 | 1.9 (0.29)
  Femoral Region 5 | 2.0 (0.32)
  Femoral Region 6 | 1.6 (0.39)
  Femoral Region 7 | 1.3 (0.25)

6. Secondary Outcome: Baseline Harris Hip Score (HHS) at Preoperative Visit
Description: The HHS is a physician tool to measure how a subject is doing following hip replacement surgery using the following scale:
  Total Scale Ranges:
  Excellent: 90 - 100 Good: 80 - 89 Fair: 70 - 79 Poor: 60 - 69 Very Poor: <60
  Subscore Ranges:
  Pain: 0 - 44 Function: 0 - 47 Absence of Deformity: 0 - 4 Range of Motion: 0 - 5
  The score ranges from 0 to 100, where, the higher the score, the better the subject outcome. Lower scores indicate a higher level of dysfunction due to hip problems.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
score on a scale
  Pain | 17.0 (7.33)
  Function | 26.0 (7.58)
  Absence of Deformity | 3.8 (0.89)
  Range of Motion | 2.7 (0.86)
  Total | 49.5 (13.53)

7. Secondary Outcome: Harris Hip Score (HHS) at 3 Month Visit
Description: as for outcome 6
Time Frame: 3 Month
Population: Overall number of participants analyzed was 20 particpants; however, for the Function and Total Overall portion of the questionnaire only 18 participants responded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
score on a scale
  Pain | 37.5 (9.56)
  Function: number analyzed (Participants) | 18
  Function | 35.1 (5.60)
  Absence of Deformity | 4.0 (0.00)
  Range of Motion | 4.1 (0.69)
  Total: number analyzed (Participants) | 18
  Total | 82.6 (10.15)

8. Secondary Outcome: Harris Hip Score (HHS) at 6 Month Visit
Description: as for outcome 6
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
score on a scale
  Pain | 40.8 (5.29)
  Function | 41.2 (5.67)
  Absence of Deformity | 4.0 (0.00)
  Range of Motion | 4.2 (0.37)
  Total | 90.1 (7.22)

9. Secondary Outcome: Harris Hip Score (HHS) at 1 Year Visit
Description: as for outcome 6
Time Frame: 1 Year
Population: Two subjects were missing results from the study site for the HHS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 17
score on a scale
  Pain | 38.0 (9.27)
  Function: number analyzed (Participants) | 15
  Function | 41.5 (7.14)
  Absence of Deformity | 4.0 (0.00)
  Range of Motion | 4.5 (0.62)
  Total: number analyzed (Participants) | 15
  Total | 87.3 (16.13)

10. Secondary Outcome: Harris Hip Score (HHS) at 2 Year Visit
Description: as for outcome 6
Time Frame: 2 Years
Population: Number of participants returning for this time point visit assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 11
score on a scale
  Pain | 40.7 (7.11)
  Function | 41.9 (5.79)
  Absence of Deformity | 4.0 (0.00)
  Range of Motion | 4.0 (0.45)
  Total | 90.6 (11.57)

11. Secondary Outcome: Harris Hip Score (HHS) at 5 Year Visit
Description: as for outcome 6
Time Frame: 5 Year
Population: Number of participants returning for this time point visit assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 9
score on a scale
  Pain | 43.6 (1.33)
  Function | 45.8 (1.48)
  Absence of Deformity | 4.0 (0.00)
  Range of Motion | 4.3 (0.50)
  Total | 97.7 (2.45)

12. Secondary Outcome: Hip Injury Osteoarthritis Outcome Score (HOOS) at Preoperative Visit
Description: The HOOS is a questionnaire that the subject completes focusing on hip pain, stiffness, and function relating to osteoarthritis of the hip. The HOOS consists of 40 items assessing 5 subscales. The 5 separate patient-relevant dimensions are Symptoms and Stiffness, Pain, Function in Daily Living, Function in Sport and Recreation, and Hip-Related Quality of Life (QoL).
  Pain includes 10 items with a total score of 0 - 100 points Symptoms includes 5 items with a total score of 0 - 100 points Function in Daily Living includes 17 items with a total score of 0 - 100 points Function in Sport and Recreation and Hip-Related QoL each include 4 items with a total score of 0 - 100 points.
  Each sub-score was transformed in a worst to best scale (0-100), where 100 indicates no symptoms and 0 indicates extreme symptoms.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
score on a scale
  Symptoms and Stiffness | 52.8 (18.53)
  Pain | 49.1 (17.50)
  Daily Living | 44.7 (17.19)
  Sports/Recreational Activities | 22.1 (19.98)
  Quality of Life | 24.7 (14.97)

13. Secondary Outcome: Hip Injury Osteoarthritis Outcome Score (HOOS) at 3 Month Visit
Description: as for outcome 12
Time Frame: 3 Months
Population: Information was not provided from the study site for two subjects in the HOOS Sports/Recreational Activities (0-100) category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
score on a scale
  Symptoms and Stiffness | 83.0 (13.42)
  Pain | 88.8 (13.39)
  Daily Living | 84.8 (12.29)
  Sports/Recreational Activities: number analyzed (Participants) | 18
  Sports/Recreational Activities | 76.0 (22.70)
  Quality of Life | 73.1 (22.86)

14. Secondary Outcome: Hip Injury Osteoarthritis Outcome Score (HOOS) at 6 Month Visit
Description: as for outcome 12
Time Frame: 6 Months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
score on a scale
  Symptoms and Stiffness | 93.0 (10.31)
  Pain | 94.2 (7.82)
  Daily Living | 93.0 (6.80)
  Sports/Recreational Activities: number analyzed (Participants) | 18
  Sports/Recreational Activities | 80.4 (17.37)
  Quality of Life | 83.8 (14.68)

15. Secondary Outcome: Hip Injury Osteoarthritis Outcome Score (HOOS) at 1 Year Visit
Description: as for outcome 12
Time Frame: 1 Year
Population: Number of participants returning for this time point visit assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 16
score on a scale
  Symptoms and Stiffness | 90.0 (14.14)
  Pain | 89.2 (14.54)
  Daily Living | 87.8 (15.62)
  Sports/Recreational Activities | 78.3 (28.8)
  Quality of Life | 82.4 (25.13)

16. Secondary Outcome: Hip Injury Osteoarthritis Outcome Score (HOOS) at 2 Year Visit
Description: as for outcome 12
Time Frame: 2 Years
Population: Number of participants returning for this time point visit assessment. Information was not provided from the study site for 1 subject in the HOOS Sports/Recreational Activities (0-100) and Quality of Life (0-100) categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 14
score on a scale
  Symptoms and Stiffness | 90.7 (8.05)
  Pain | 92.5 (10.28)
  Daily Living | 89.9 (12.54)
  Sports/Recreational Activities: number analyzed (Participants) | 13
  Sports/Recreational Activities | 81.6 (20.60)
  Quality of Life: number analyzed (Participants) | 13
  Quality of Life | 81.7 (22.74)

17. Secondary Outcome: Hip Injury Osteoarthritis Outcome Score (HOOS) at 5 Year Visit
Description: as for outcome 12
Time Frame: 5 Years
Population: Information was not provided from the study site for 1 subject in the HOOS Pain (0-100), Daily Living (0-100), Sports/Recreational Activities (0-100), and Quality of Life (0-100) categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIS Stem
Number analyzed (Participants) | 10
score on a scale
  Symptoms and Stiffness | 96.5 (6.69)
  Pain: number analyzed (Participants) | 9
  Pain | 98.3 (4.15)
  Daily Living: number analyzed (Participants) | 9
  Daily Living | 97.2 (5.27)
  Sports/Recreational Activities: number analyzed (Participants) | 9
  Sports/Recreational Activities | 85.6 (21.91)
  Quality of Life: number analyzed (Participants) | 9
  Quality of Life | 95.8 (6.99)

18. Secondary Outcome: Radiographic Assessment at Preoperative Visit (Yes/No Components)
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view. The span of the bone-prosthesis interface for each component was broken down into zone systems. The scoring system was based on the measurement of radiolucent lines (in millimeters) in each zone. The checklist reviewed radiolucencies, migration, osteolysis, and stress shielding.
  The Brooker Classification was defined as:
  Class 0 - absence of radiographic heterotopic ossification Class 1 - islands of bone within soft tissues Class 2 - bone spurs originating from pelvis or proximal end of femur with at least 1 cm between opposing bone surfaces Class 3 - bone spurs originating from pelvis or proximal end of femur reduced to <1 cm Class 4 - apparent bone ankyloses of the hip
Time Frame: Discharge
Measure: Count of Participants; unit: Participants
Groups:
- MIS Stem: Patients with non-inflammatory and inflammatory degenerative joint disease (DJD) who required a primary total hip replacement (THR) and had the MIS femoral stem/modular neck implanted. There was no assignment of study treatment: all subjects had implantation of the MIS femoral stem/modular neck during THA.
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
Participants
  No Problems on Checklist: Yes | 20
  No Problems on Checklist: No | 0
  Acetabular Component Position Degree: Yes | 0
  Acetabular Component Position Degree: No | 20
  Stem Subsidence: Yes | 0
  Stem Subsidence: No | 20
  Evidence of Acetabular Component Failure: Yes | 0
  Evidence of Acetabular Component Failure: No | 20
  Evidence of Femoral Component Failure: Yes | 0
  Evidence of Femoral Component Failure: No | 20
  Brooker Classification: Yes | 0
  Brooker Classification: No | 20

19. Secondary Outcome: Radiographic Assessment at 3 Month Visit (Yes/No Components)
Description: as for outcome 18
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
Participants
  No Problems on Checklist: Yes | 20
  No Problems on Checklist: No | 0
  Acetabular Component Position Degree: Yes | 0
  Acetabular Component Position Degree: No | 20
  Stem Subsidence: Yes | 0
  Stem Subsidence: No | 20
  Evidence of Acetabular Component Failure: Yes | 0
  Evidence of Acetabular Component Failure: No | 20
  Evidence of Femoral Component Failure: Yes | 0
  Evidence of Femoral Component Failure: No | 20
  Brooker Classification: Yes | 0
  Brooker Classification: No | 20

20. Secondary Outcome: Radiographic Assessment at 1 Year Visit (Yes/No Components)
Description: as for outcome 18
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
Participants
  No Problems on Checklist: Yes | 19
  No Problems on Checklist: No | 1
  Acetabular Component Position Degree: Yes | 0
  Acetabular Component Position Degree: No | 20
  Stem Subsidence: Yes | 1
  Stem Subsidence: No | 19
  Evidence of Acetabular Component Failure: Yes | 0
  Evidence of Acetabular Component Failure: No | 20
  Evidence of Femoral Component Failure: Yes | 0
  Evidence of Femoral Component Failure: No | 20
  Brooker Classification: Yes | 0
  Brooker Classification: No | 20

21. Secondary Outcome: Radiographic Assessment at 5 Year Visit (Yes/No Components)
Description: as for outcome 18
Time Frame: 5 Year
Population: All participants available at this time point visit assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Stem
Number analyzed (Participants) | 10
Participants
  No Problems on Checklist: Yes | 10
  No Problems on Checklist: No | 0
  Acetabular Component Position Degree: Yes | 0
  Acetabular Component Position Degree: No | 10
  Stem Subsidence: Yes | 0
  Stem Subsidence: No | 10
  Evidence of Acetabular Component Failure: Yes | 0
  Evidence of Acetabular Component Failure: No | 10
  Evidence of Femoral Component Failure: Yes | 0
  Evidence of Femoral Component Failure: No | 10
  Brooker Classification: Yes | 0
  Brooker Classification: No | 10

22. Secondary Outcome: Radiographic Assessment at Discharge Visit
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: Discharge
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
degree
  Femoral Valgus Position Degree | 0 (0)
  Acetabular Component Position Degree | 40.9 (3.44)

23. Secondary Outcome: Radiographic Assessment at 3 Month Visit
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
degree
  Femoral Valgus Position Degree | 0 (0)
  Acetabular Component Position Degree | 41.3 (2.90)

24. Secondary Outcome: Radiographic Assessment at 1 Year Visit
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
degree
  Femoral Valgus Position Degree | 0 (0)
  Acetabular Component Position Degree | 41.3 (2.90)

25. Secondary Outcome: Radiographic Assessment at 5 Year Visit
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 5 Year
Population: All available subjects participating in this time point visit assessment.
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
degree
  Femoral Valgus Position Degree: number analyzed (Participants) | 10
  Femoral Valgus Position Degree | 10.5 (2.12)
  Acetabular Component Position Degree | 40.6 (3.41)

26. Secondary Outcome: Radiographic Assessment at Discharge Visit (Neutral/Valgus Component)
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: Discharge
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
Participants
  Neutral | 20
  Valgus | 0

27. Secondary Outcome: Radiographic Assessment at 3 Month Visit (Neutral/Valgus Component)
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
Participants
  Neutral | 20
  Valgus | 0

28. Secondary Outcome: Radiographic Assessment at 1 Year Visit (Neutral/Valgus Component)
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Stem
Number analyzed (Participants) | 20
Participants
  Neutral | 20
  Valgus | 0

29. Secondary Outcome: Radiographic Assessment at 5 Year Visit (Neutral/Valgus Component)
Description: Radiographs were obtained from the anteroposterior (AP) view as well as the lateral view.
Time Frame: 5 Years
Population: All available subjects participating in this time point visit assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | MIS Stem
Number analyzed (Participants) | 10
Participants
  Neutral | 8
  Valgus | 2

ADVERSE EVENTS:
Time Frame: The time frame for collection of AEs is from the signing of the Informed Consent through Study Exit, an average of 5 years.
Description: Device-related adverse events are defined as any of the following: any device implant component failure including any of the following exact or similar descriptive nomenclature: a) revision, fracture, crack, chip, flake, split, splinter, shatter, break, or wear-through; b) device wear particle induced osteolysis, inflammation, etc. (wear debris may be metal and/or UHMWPE in composition); and c) any device component experiencing dislocation, subluxation, subsidence, migration, or loosening.
Arm/Group | MIS Stem
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIS Stem (N=20)
Death (General disorders) | 2 (2) — Death from unknown causes
Atrial fibrillation (Congenital, familial and genetic disorders) | 1 (1)
Cut hand - hospital admission for intervenous (IV) antibiotics (Injury, poisoning and procedural complications) | 1 (1)
Contralateral THR secondary to osteoarthritis (OA) (Musculoskeletal and connective tissue disorders) | 2 (2)
Unicompartmental knee replacement secondary to OA (Musculoskeletal and connective tissue disorders) | 2 (3)
Cholecystectomy (Gastrointestinal disorders) | 1 (1)
Alzheimer's Disease (Nervous system disorders) | 1 (1)
Subsidence of femoral prosthesis; revision in THR (Product Issues) | 1 (1)
Dislocation THR (Product Issues) | 1 (2)
Bleeding gastric ulcer (Gastrointestinal disorders) | 1 (1)
Osteolysis region 1, 3-7 on radiograph (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain on weight-bearing lower thigh (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIS Stem (N=20)
Paroxysmal Atrial fibrillation (Cardiac disorders) | 1 (1)
Cortical thickening region 3 (Musculoskeletal and connective tissue disorders) | 11 (11)
Newly diagnosed hypoparathyroidism (Metabolism and nutrition disorders) | 1 (1)
Mild sclerosis over weight-bearing aspect of acetabulum on x-ray (Musculoskeletal and connective tissue disorders) | 1 (1)
Adductor tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sprained Adductors (Injury, poisoning and procedural complications) | 1 (1)
Thigh and trochanteric pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Condensation around tip of stem on x-ray femur (Musculoskeletal and connective tissue disorders) | 1 (1)
Trochanteric pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There was a decreased compliance rate at the 3 year follow-up and a 50% termination rate by the 5 year follow-up resulting in a much smaller sample sizes for data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less